CLINICAL TRIAL: NCT07194759
Title: Patient and Family Health Literacy - a Survey Among 5000 People
Brief Title: Health Literacy Levels of Patients Living With Type 2 Diabetes and Multi-disease and Their Families Using HLQTM
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-MS-1-2025
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Health Literacy
Keywords: Diabetes Mellitus; Outpatients; Socioeconomic factors; Multiple chronic conditions; Family
MeSH Terms: conditions — Diabetes Mellitus; Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify health literacy strengths and needs among people living with type 2 diabetes and multi-disease and their family members.

DETAILED DESCRIPTION:
Living with diabetes and multi-disease affects not only the individual but also the social network around the person, as self-management is dependent on the ability to change one's lifestyle and manage the consequences of disease. In other words, health literacy strengths and needs of the individual and family members are determinants of how people manage living with type 2 diabetes. Thus, we hypothesise that diabetes management is influenced by the patient's and family members' health literacy. Knowledge about their health literacy could further enhance a patient- and family-centred approach to diabetes treatment and care, improving self-management and promoting health.

ELIGIBILITY:
Inclusion Criteria:

* living with Type 2 diabetes and multi-disease
* cognitively able to participate
* following an outpatient care program

Exclusion Criteria:

* patients in palliative care
* inability to read or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients and/or family members from four university hospitals in the Region of Southern Denmark. The patients will be invited to participate when they receive a questionnaire. This questionnaire is designed to provide participant information and consent prior to the sociodemographic questions and the health literacy questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Health Literacy Questionnaire (HLQ) | At Enrollment
  The Health Literacy Questionnaire (HLQ) is a 44-item validated questionnaire on health literacy. It consists of two parts, one part with 23 questions answered with a 4-point Likert Scale (strongly disagree = 1, disagree = 2, agree = 3, and strongly agree = 4). The second part has 21 questions answered with a 5-point Likert Scale (can't do/always difficult = 1, usually difficult = 2, sometimes difficult = 3, usually easy = 4, always easy = 5). The patient must select one of the scales for each of the 44 questions.
  The answers are self-reported via REDCap, one time after the survey is distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Frans Brandt Kristensen, Study Chair — University Hospital of Southern Denmark, Hospital Sønderjylland
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No